CLINICAL TRIAL: NCT05537727
Title: Robotic Minimally Invasive Gynecological, Urological, and General Surgery With Dexter
Brief Title: Robotic MIS With Dexter
Status: Completed | Type: Observational
Sponsor: Distalmotion SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-01
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hysterectomy; Partial Nephrectomy; Right Colectomy
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: robotic-assisted surgery — Gynecology: robot-assisted and laparoscopic hysterectomy for benign or low risk malignant disease
Device: robotic-assisted surgery — Urology: robot-assisted and laparoscopic partial nephrectomy
Device: robotic-assisted surgery — General surgery: robot-assisted and laparoscopic right colectomy

SUMMARY:
The purpose of this study is to confirm the perioperative and early postoperative safety and clinical performance of the Dexter Robotic System (Dexter Surgical System, Model DM-L6).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Patient agrees to perform the 30-day follow-up assessment
* Able to provide signed Informed Consent, according to local regulation

Exclusion Criteria:

* Morbidly obese patients.
* Any and all relative and absolute contraindications to endoscopic surgical technique applicable to the use of conventional endoscopic surgical instruments.
* Bleeding diathesis.
* Pregnancy.
* Patients with pacemakers or internal defibrillators.
* Any planned concomitant procedures.
* Patient deprived of liberty by administrative or judicial decision or under legal guardianship.
* Participation in another interventional clinical trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of the modified intent-to-treat (mITT) sample. This is defined as the set of patients who were enrolled in the trial and on whom robotic-assisted surgery with Dexter was at least started.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
occurrence of serious (Clavien - Dindo grades III-V), device related adverse events. | perioperatively up to 30 days
successful completion of the Dexter-assisted procedure, i.e. free of any device related permanent conversion to an open or fully laparoscopic surgical approach. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hahnloser, MD, Principal Investigator — CHUV
Locations (5):
- France (2):
  - Hopital Paris Saint-Joseph, Paris
  - Centre Hospitalier de Saintes, Saintes
- UKSH, Kiel, Germany
- Switzerland (2):
  - Inselspital, Bern
  - CHUV, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided